CLINICAL TRIAL: NCT05165446
Title: Novel MRE Technique to Assess Tissue Viscoelasticity as a Risk Factor for Liver Cancer
Brief Title: Novel MRE Technique to Assess a Risk Factor for Liver Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Natalie Torok (Other)
Responsible Party: Sponsor-Investigator, Natalie Torok, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 62249
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Fatty Liver; NAFLD; Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 tablespoon (13 mL) blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this proposal is to investigate a novel imaging method to identify patients with non-alcoholic steatohepatitis (NASH) who are at risk for hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
NASH is the most common cause of chronic liver disease, and it is estimated that 40-50% of patients with obesity and T2DM have NASH. NASH can lead to HCC with the risk increasing 2-3 fold in patient with poor glycemic control. Unless caught early, HCC has a poor prognosis with no effective therapies. A unique feature of HCC in NASH is that it often arises at a pre-cirrhotic stage, and the prognosis is often dismal. There are no current surveillance strategies for these pre-cirrhotic patients. Based on our animal models and pilot patient studies, we developed a novel paradigm that linked liver matrix changes to a more aggressive HCC phenotype. Our goal is to develop an imaging-based surveillance tool that will identify early matrix changes that may predispose to HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant/non-lactating women ≥ 18 years of age
2. Diagnosis of NASH
3. Diagnosis of pre-cirrhotic fibrosis (F1-F3), diagnosed as per standard of care (history, exam, laboratory tests, Fibroscan, within 6 months of enrollment)
4. Na-MELD < 9: The Na-MELD (sodium-Model for End Stage Liver Disease) score is routinely used to assess liver synthetic function and life expectancy. Patients with Na-MELD<9 have less than 1.9% 3 months liver-related mortality risk, and their liver synthetic function is normal.
5. Groups both with and without T2DM will be enrolled.
6. Women of childbearing potential must agree to at least two methods of contraception.
7. Will not participate in any other clinical trial for the duration of the study
8. Will not consume alcohol for the duration of the study
9. If on vitamin E, pioglitazone or any anti diabetic treatment prior to the study, will have been on stable therapies for 6 months prior to enrolment.
10. Able to undergo 3 Tesla MRI and complete MRI screening form
11. Ability to understand and the willingness to sign a written informed consent document.
12. ECOG or Karnofsky Performance Status will be not be employed

Exclusion Criteria:

1. Presence of any other form of liver disease, including viral hepatitis, autoimmune hepatitis, alcoholic liver disease, genetic causes of chronic liver disease, cardiogenic liver disease, and HIV positivity (can cause liver fibrosis).
2. ALT>300 U/l
3. Total serum bilirubin ≥ to 1.3 mg/dL (Gilbert's Syndrome patients are excepted)
4. International Normalized Ratio (INR) ≥ 1.3
5. MELD>9
6. Serum creatinine >2.0mg/dl
7. Known alcohol abuse or alcohol use disorder (AUDIT profile and/or pos. urine ethylglucuronide):

   * >20 g/day for women
   * >30 g/day for men
8. Active substance abuse
9. Platelet count ≤100//mm3
10. Hemoglobin <11 g/dl in females or <12 g/dl in males
11. Presence/history of HCC, or other primary or metastatic cancer to the liver.
12. History of liver transplantation
13. History of bariatric surgery
14. History of inflammatory bowel disease
15. History of advanced pulmonary disease
16. Any concerns regarding compliance by enrolling physician
17. Pregnant or lactating women.
18. Presence of cardiac implantable electronic device (CIED)
19. History of CIED with retained leads
20. Presence of any metallic foreign body that is unsafe for the MRI environment
21. Inability to undergo MRI based on responses to the MRI screening form
22. History of claustrophobia or the need for sedation to undergo MRI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include one group of healthy subjects and two groups with 15 patients each which will enroll in parallel, one group with type 2 diabetes mellitus (T2DM), and one group without DM.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Novel MRE technique to assess tissue viscoelasticity as a risk factor for liver cancer | For individual patients: duration of the study 8 weeks (including lab, scheduling the MR and 4w post MR period).
  Safety:MRE evaluation of the liver for stiffness is a standard of care test. We do not expect issues as this is a non-invasive technique. Our MR may require a longer session compared to the traditional MRE (40 minutes of scan time for multifrequency MRE, as compared to 25 minutes for conventional MRE). However, all issues, patient symptoms will be recorded.
  Technical Feasibility: The MRE algorithm we will use has previously been shown to produce data from a different scanner platform, across all frequencies. Feasibility of multifrequency MRE will be assessed by descriptive summary of technical success and image quality for each of the individual reconstructed MRE datasets (stiffness, elasticity, and viscosity). Mean and standard deviation for the MRE outcome variables viscosity elasticity and stiffness will be presented and tested for the difference in means between the 2 groups by way of ANOVA, and if a difference is found, followed by Tukey's test.

SECONDARY OUTCOMES:
Studies on liver injury and glycemic control. | For individual patients: duration of the study 8 weeks
  assess correlation to liver injury (AST, ALT) assess correlation to glycemic control HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Torok, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Stanford, California, United States